CLINICAL TRIAL: NCT00374023
Title: A Study on Immunological Effect of Vitamin A and Zinc in a Placebo Controlled 4 Cell Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 93-012
Record Dates: First submitted 2006-09-07; First posted 2006-09-08 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 1993-05

CONDITIONS: Immunity; Diarrhea; Respiratory Tract Infections
Keywords: Zinc; vitamin A; immunity; morbidity; height gain; weight gain; Children aged between 1 and 3 years; Weight for age between 70% and 61% of NCHS standard; Acute diarrhoeal Patients; No signs of vitamin A deficiency; Who has not received measles vaccine
MeSH Terms: conditions — Diarrhea; Respiratory Tract Infections; Weight Gain | interventions — Zinc; Vitamin A

INTERVENTIONS:
Drug: Zinc, or Vitamin A or both

SUMMARY:
Vitamin A deficiency in children is associated with increased mortality and morbidity due to respiratory tract and diarrhoeal infections. Vitamin A supplementation has been shown in some studies to reduce morbidity due to respiratory diseases. However, other studies to reduce could not document such benefit from vitamin A supplementation. The role of vitamin A on immunity in humans is not yet clear due to inconclusive results. To evaluate immune changes and compare those with of a known immunopotent agent like zinc, a randomised double blind study will be carried out in 1-3 year aged children without acute illness and wt/age between 61% and 70% of NCHS standard. Baseline anthropometry and vitamin A status will be determined using MRDR test and immune status will be estimated. Each group consisting of 50 children will either receive vitamin A 200,000 IU over 7 days or 40 m elemental zinc daily for 7 days or both or placebo. After 8 weeks immunity test will be repeated. Immunity tests will include serum 1gA, 1gM, 1gG an lymphocyte simulation and 8 antigen multiple skin test. Undiminished children will be given measles vaccine and serum titre will be measured before and after supplementation. Vitamin A status will be estimated by MRDR test. Vitamin A2 will be given and 1ml blood sample will be collected after 5 hours to see the ratio of vitamin A1 and A2 (<0.06 as cut off) as the modified relative dose response (MRDR test). Doses of vitamin A or zinc will be repeated at the completion of 2 month. The results will be compared between groups and within groups at baseline and after 6 weeks. The study will generate information which will help to examine the immune response of vitamin A therapy in children as an underlying factor for reduction in mortality or morbidity. The study will be completed within a year.

DETAILED DESCRIPTION:
Immunological indicators will be monitored at the beginning and after 8 weeks of giving vitamin A or zinc in a double blind randomized trial. A clinical based study will be done to see the effect of zinc or vitamin A supplementation in malnourished subjects. Vitamin A status will be estimated using the newer indicator, modified relatively dose response. (MRDR).Procedure:Study population:Children aged 1 to 3 years will be included. Forty children in each group will be assigned to either group A group B and group C and group D. children will be selected from families within Dhaka city who come to the diarrhoea treatment centre of ICDDR,B.Inclusion criteria:1. Children aged between 1 and 3 years having weight for age between 70% and 61% of NCHS standard.2. Who come to the out patient department of ICDDR,B for treatment of acute water diarrhoea with3. No signs of vitamin A deficiency (non invasive diarrhoea and without systematic infection) and has not received vitamin A during last 4 months.4. Who has not received measles vaccine and did not have measles primarily identified for the study.5. Children who has not reside in and around Dhaka city After one week recovery from diarrhoea:1. Baseline immunological profile will be studied.2. Intervention for one week at the schedule doses and immunological profile will be repeated after 8 weeks.Study groups are:A. Zinc B. Vitamin A C. Zinc and vitamin A D. PlaceboExclusion criteria:1. Children who needs immediate vitamin A supplementation (clear sign of vitamin deficiency)2. Children who received vitamin A within the last 4 months3. Children with other systematic infection4. Subjects who develop any kind of sign and symptoms of vitamin A deficiency will be given vitamin A and will be analysed separately.Randomisation procedure: Parents who give their consent for the study will be selected. Children will be randomised into four groups to receive either of the treatments. A master randomisation chart will be prepared using table in permuted block design by dividing serial number into four equal groups. There will be no need for stratification but according to the selection criteria, better nourished (70% wt/age) or severely malnourished (60%) children will be excluded. Severely malnourished patients with diarrhoea may immediately need vitamin A or well nourished will not show effect of supplements. Steps will be kept to compensate dropouts.The intervention and non-intervention groups will receive identical bottles and syrups with some flavour and only single unique serial number will be written outside the bottles. The number will indicate an exact subject of study and will be kept out of the reach of the investigators. The children will receive the 2nd dose at 8 weeks with vitamin A or zinc who has not received that in the first dose without breaking the randomization code. The code will be broken only after completion of study and analysis according to groups.Base line survey will be done to take socio-economic information, dietary habits, previous illness, immunization, washing of hands and water use, frequency of cooking of food containing vit A, cooking method, and frequency of use of green leafy vegetables.In the beginning of the study, baseline vitamin A status will be determined using MRDR test. Anthropometry will be done to select children at the baseline, at the end of 8 weeks, and subsequent months for 6 months. Duration, frequency, dose:One teaspoonful, (5 ml) syrup will be given in a twice-daily schedule for 7 days.Composition of syrup:For all groups, the main vehicle and bulk of the base syrup will consist of the same chemicals; in addition to this, each group will have either of the treatment substance (i.e. zinc or vitamin A or both or none).Syrup A : Quantity per 5 ml Zinc acetate 20 mg elemental

Syrup B :

Vitamin A palmitate 15,000IU

Syrup C :

Zinc : 20 mg elemental + vitamin A : 15,000 IU Syrup D : Y base substance Base substance: Ascorbic acid 30 mg Glycerine USP 1.2 ml Propylene glycol USP 0.75 ml Sorbitol 70 % BP 2.0 ml Methyl Paraban USFN 3.5 mg Polysorbate-80 50 mg (Tween-80) BPC Lemon oil pH grade 0.0125 ml Caramel Brown colour 1 mg Powder water 0.75 ml Organization of the study:The study will be conducted among the children who will attend the out patient department of the clinical research centre of ICDDR,B. Children will be selected at the acute diarrhoea phase who will attend only with non invasive simple or mild diarrhoea within the nutritional status defined earlier of NCHS standard. The children will be taken for study 1 week after the recovery of diarrhoea and the first immunological test at base line will be done at this time. Mothers will be instructed on the dose. A twice-daily dose of syrup for one week will be schedule for better compliance of the children. After completion of doses at 8 weeks, the immunity test will be repeated a 8 weeks. Tears will be collected in a small piece of sponge and will be used for secretary 1 gA estimation. Skin test for Cell Medicated Immunity will be performed in each child regardless of treatment group with multitest kit developed by Institute Merieux. These children will be followed up every alternate day for the 1st week and then weekly for development of any illness for 2 months. Necessary treatment measures will be undertaken.Clinical care: Patient care will be provided on clinical problems identified during treatment of diarrhoea or follow up. A team of medical officers and paramedics will examine and record the vitamin A deficiency symptoms and other medical problems on a predesigned questionnaire and provide the necessary care. Any children develop an acute symptom of night blindness or Bitot's spot will be given a vitamin A capsule (200,000 in) which will be recorded.Baseline test on immunity will be performed by the following tests:Components of immunity and other variables:1. Eight antigens multiple skin tests measured by 48 hours.2. Eight 1gA, 1gM3. MRDR, plasma 1gA, 1gM, 1gG.(This will require 2 ml blood)4. Lymphocyte proliferation assays.For T lymphocytes- PHA, Con A antigen will be used For T and B lymphocytes - PWM (Poke weed Mitogen)(This will require 3 ml blood in heparinized tube) 5. Lymphocyte Phenotype using monoclonal antibodies to CD3, CD4, CD8, CD20.Schedules: for immunity test, skin test before dose and after 8 weeks. MRDR will be done at base line and at 8 weeks.6. Base line titre of measles antibody 1gG will be measured and will be followed by a dose of measles vaccine and titre be measure at 8 weeks of supplementation.7. 'Serum zinc, RBP, albumin & alkaline phosphatase at baseline after 8 week.Anthropometry will be done with weight, height, MUAC, at base line, at 8 weeks.Body weight- will be measured (nude) with an electronic scale with a 1gLength:- will be measured in knee-heel vernier with 1mm sensitivity. Data collection on morbidityA predesigned questionnaire will be used to record incidence and duration of illness during the follow up period

ELIGIBILITY:
Inclusion Criteria:

1. Children aged between 1 and 3 years having weight for age between 70% and 61% of NCHS standard.
2. Who come to the out patient department of ICDDR,B for treatment of acute water diarrhoea with
3. No signs of vitamin A deficiency (non invasive diarrhoea and without systematic infection) and has not received vitamin A during last 4 months.
4. Who has not received measles vaccine and did not have measles primarily identified for the study.
5. Children who has not reside in and around Dhaka city

Exclusion Criteria:

1. Children who needs immediate vitamin A supplementation (clear sign of vitamin deficiency)
2. Children who received vitamin A within the last 4 months
3. Children with other systematic infection
4. Subjects who develop any kind of sign and symptoms of vitamin A deficiency will be given vitamin A and will be analysed separately

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 147
Dates: Start 1993-07-01; Primary Completion 1995-11-30 (Actual); Study Completion 1995-11-30 (Actual)

PRIMARY OUTCOMES:
Immunization test result - IgA(tears, T-lymphocyte number, Proportion, Phenotype, CD4%. CD8%, CD20% PHA, CON-A, PWM at baseline and after 6 weeks.
Skin test CM1
MUAC
Height

SECONDARY OUTCOMES:
Morbidity: new attacks of respiratory infection + duration of respiratory infection
Attacks of diarrhoea and duration
Fever without respiratory infection

CONTACTS AND LOCATIONS:
Overall Officials: Swapan K Roy, MBBS, PhD, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- Dhaka Hospital, ICDDR,B, Dhaka, Bangladesh

REFERENCES:
- [Derived] Imdad A, Rogner J, Sherwani RN, Sidhu J, Regan A, Haykal MR, Tsistinas O, Smith A, Chan XHS, Mayo-Wilson E, Bhutta ZA. Zinc supplementation for preventing mortality, morbidity, and growth failure in children aged 6 months to 12 years. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD009384. doi: 10.1002/14651858.CD009384.pub3. PMID 36994923